CLINICAL TRIAL: NCT02051127
Title: Sustainable Working Life With Reduced Stress Levels - The Effects of Physical Training on Physiological and Psychological Stress-reactions and Cognitive Function.
Brief Title: The Effects of Physical Training on Physiological and Psychological Stress-reactions and Cognitive Function.
Acronym: ASTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ISM-01-2013; 2012-0484 (Other Grant/Funding Number: FORTE)
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Healthy Volunteers; Sedentary Lifestyle
Keywords: Exercise; Physical Fitness; Stress, Psychological; Cognition; Psychophysiology; Ergometry; Exercise Test; Sedentary Lifestyle
MeSH Terms: conditions — Sedentary Behavior; Motor Activity; Stress, Psychological | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Physical training Duration: 45-60 minutes Frequency: 3 times per week Intensity: mean heart rate > 75% of maximum heart rate determined by exercise test before start of the intervention
  Interventions: Other: Exercise
- Control (No Intervention): Instructed to continue with their sedentary behavior for another 6 months.

INTERVENTIONS:
Other: Exercise — Physical training Duration: 45-60 minutes Frequency: 3 times per week Intensity: mean heart rate > 75% of maximum heart rate determined by exercise test before start of the intervention
  Arms: Exercise

SUMMARY:
One of the biggest challenges of today is the high stress levels among employees in companies and organizations. Physical exercise may be an effective preventive measure for stress-related problems. This relatively simple and inexpensive action is believed to be important for increasing and maintaining work ability and reduce the cost of stress-related ill health in the workplace.

The aim is to investigate how regular physical exercise affects the individual's ability to mentally and physiologically cope with stress. Acute stress physiological responses are measured before and after a 6 -month intervention, where 100 untrained individuals are randomized to either regular physical exercise or a control group.

The hypothesis is that exercise leads to lesser activation of the individual's stress physiological systems and to an efficient physiological protection system. Mental ability to handle stress is also studied as well as possible effects on the brain's cognitive functions. From a work perspective, cognitive impairment due to high exposure to stress is a major problem leading to substantial costs in businesses and organizations as a result of reduced performance and production.

We believe that physical activity can alter and mitigate individual stress reactions. This study brings new knowledge that can contribute to increased motivation to prioritize physical activity in everyday life. The study could also provide evidence for businesses and organizations of the benefits of engaging in interventions and fitness initiatives to facilitate/enable increased physical activity in daily life for its employees. With an aging population, we are expected to work longer, which poses a challenge as the ability to manage stress and maintain cognitive abilities decline with age. For older employees, regular physical activity could be an important factor directly affecting the prospects for a sustainable working life.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported good health
* Sedentary
* Work or study at least 50%

Exclusion Criteria:

* Diabetes
* Cardiovascular disease
* Blood pressure > 140/90
* Psychiatric disease
* Anemia
* Medication with substances that could affect any of the outcome measures

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2017-04-03 (Actual)

PRIMARY OUTCOMES:
Cortisol responses to acute psychosocial stress. | 6 months after start of intervention
  Serum cortisol (nmol/l) profile after exposure to the Trier Social Stress Test (TSST).

SECONDARY OUTCOMES:
Cognitive function | 6 months after start of intervention
  Performance of the CNS Vital Signs (CNSVS) cognitive test battery.
Self-reported stress sensitivity and symptoms | 6 and 12 months after start of intervention
  Assessed with the Perceived Stress Scale (PSS), Coping Inventory for Stressful Situations (CISS), Shirom Melamed Burnout questionnaire (SMBQ), Hospital Anxiety and Depression scale (HAD) and Patient Health Questionnaire (PHQ-15).
Adrenocorticotropic hormone (ACTH) response to psychosocial stress | 6 months after start of intervention
  ACTH in plasma (pmol/L) after exposure to the TSST
Dehydroepiandrostreone (DHEA) and dehydroepiandrosterone sulfate (DHEAS) response to psychosocial stress | 6 months after start of the intervention
  DHEA(S) in serum (µmol/L) after exposure to the TSST

OTHER OUTCOMES:
Autonomic responses to acute psychosocial stress | 6 months after start of intervention
  Heart rate and blood pressure during and after the Trier Social Stress Test (TSST).
Neuroendocrine and autonomic responses to exercise test | 6 months after start of intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ingibjörg H Jonsdottir, Professor, Principal Investigator — Västra Götalandsregionen
Locations (1):
- The Institute of Stress Medicine, Gothenburg, VGR, Sweden

REFERENCES:
- [Derived] Arvidson E, Dahlman AS, Borjesson M, Gullstrand L, Jonsdottir IH. The effects of exercise training on hypothalamic-pituitary-adrenal axis reactivity and autonomic response to acute stress-a randomized controlled study. Trials. 2020 Oct 27;21(1):888. doi: 10.1186/s13063-020-04803-3. PMID 33109273
- See also: Webpage of the Institute of Stress Medicine — http://www.vgregion.se/stressmedicin